CLINICAL TRIAL: NCT06118554
Title: 3D Printing for Topical Nasal Corticosteroid Irrigations: a Randomized Clinical Trial.
Brief Title: 3D Printing to Improve Nasal Irrigation Outcome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kai Zhao, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020H0068
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Chronic Rhinosinusitis Without Nasal Polyps
Keywords: 3D modeling

STUDY DESIGN:
Intervention Model Description: All patients were prescribed an 8-week course of daily 2 mg of mometasone irrigation (Advanced Rx Compounding Pharmacy, Fort Washington, Pennsylvania) using 240 mL Sinus Rinse bottles (NeilMed Pharmaceuticals Inc, Santa Rosa, CA). The control group (CG) irrigated in the standard FDA consumer-recommended position, defined as leaning forward with a natural ear-to-shoulder head tilt. Backfill group (BG) subjects irrigated with a head tilt of 90 degrees ear-to-shoulder and used the nostril closest to the ground. Finally, the model group (MG) irrigated in an optimal position based on their 3D nasal replica. This patient-specific position was communicated to each MG patient with clear instructions during an in-person training session. All patients were required to record their daily compliance, if they changed head position, and what head position they changed to during the course of the treatment.
Who Masked: Care Provider, Investigator
Masking Description: The study was single-blinded as the MG patients unavoidably knew of their experimental group assignment due to the provided 3D-printed nasal model. However, patients in BG and CG were not told the existence of other groups. Clinical providers were blinded to the patients' assigned group when assessing clinical outcomes and Lund-Mackay score, and the principal investigator was blinded to the patients' clinical outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control group (Active Comparator): The control group (CG) irrigated in the standard FDA consumer-recommended position, defined as leaning forward with a natural ear-to-shoulder head tilt.
  Interventions: Other: Irrigation head position
- Backfill group (Experimental): Backfill group (BG) subjects irrigated with a head tilt of 90 degrees ear-to-shoulder and used the nostril closest to the ground.
  Interventions: Other: Irrigation head position
- Model group (Experimental): Finally, the model group (MG) irrigated in an optimal position based on their 3D nasal replica. This patient-specific position was communicated to each MG patient with clear instructions during an in-person training session.
  Interventions: Other: Irrigation head position

INTERVENTIONS:
Other: Irrigation head position — Patients irrigated their sinuses with once daily 2 mg mometasone using 240 mL NeilMed sinus rinse bottles for 8 weeks. The only factor that varied between groups was the head position patients irrigated in.

SUMMARY:
Three-dimensional (3D) printing has been an emerging technology with uses in a wide array of fields. This research aims to use 3D printing as a tool to provide personalized education to maximize treatment efficacy based on the patient's individual anatomy. With increased irrigation to the sinuses, we hypothesize there will be improved patient satisfaction and higher quality of life. The outcomes of this research could lead to a new option for patients who live with chronic rhinosinusitis are not candidates for surgery or are interested in less invasive options. The 3D printed nasal replica is not something that would be implanted, rather it is a hand-held device used specifically for participants to better understand their nasal anatomy.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is one of the most common medical conditions in the US, affecting an estimated 13% of adults, or some 30 million people. It accounts for 12.5 million physician office visits each year and an annual health care expenditure of $5.8 billion (National Health Interview Survey 2009, CDC). Major symptoms include nasal obstruction, facial pain/pressure, nasal discharge, purulence in the nasal cavity, and loss of smell. These symptoms significantly impact patient quality of life, even compared to chronic debilitating diseases such as diabetes and congestive heart failure.

Topical therapies play an integral role in the management of CRS, and high-volume irrigation delivery (e.g., neti pot, squeeze bottles) is more effective for achieving distribution to the sinuses than other topical delivery methods such as nasal sprays, nebulizers, or atomizers. Saline irrigations have been recommended in a number of clinical scenarios, including initial management of CRS and postoperative care. High-volume irrigations have also shown benefits for medication delivery, such as with mupirocin and corticosteroids. However, due to the intricate and variable anatomy of the human nasal airway, the efficacy of topical irrigations is inconsistent and difficult to predict. Previous studies from our group and others have shown that nasal irrigant may not reliably penetrate all sinuses, and the effectiveness varies depending on specific sinuses, head positions, injection angle, pressure, flow rates, and other factors. We currently do not have a clear understanding of the optimal delivery technique(s). In efforts to improve these outcomes, the efficacy of topical irrigation delivery to target sinuses is an area of active research. Yet, investigations have been limited by labor-intensive methodologies, such as cadaver studies or using colored dyes followed by endoscopy to visualize where the irrigation might have reached. Other studies have used irrigations with iodinated contrast followed by computed tomography (CT) scans to determine which sinuses collect contrast material. Similarly, technetium 99m sulfur colloid and fluorescein have also been used as tracers to visualize the distribution of sinus irrigations. These labor-intensive techniques are difficult to apply to a large sample size. They increase patient risk and commonly capture only where the irrigation fluid has been at the end of irrigation, but not the details of irrigation flow paths that would allow us to understand why the irrigation outcomes vary.

From both patients' and clinicians' perspectives, the lack of clear prediction of patient-specific irrigation outcomes can be frustrating, as clinicians prescribe a rigorous daily irrigation routine but have no assurance that what patients are doing is effective. When symptoms fail to improve after courses of irrigation, it is difficult to determine whether the added medication is not working, or the irrigation does not reach clinically relevant targets deep within the sinuses. Many patients and surgeons thus opt for systemic medication or surgery, which increases risk of overmedication, growth of resistant organisms, systemic side effects, and serious risk from surgery.

The purpose of this study was to propose a novel idea: applying three-dimensional (3D)-printing technology based on individual patients' computed tomography (CT) scans to determine an optimal personalized nasal irrigation strategy (head positions, angle of injection, flow rates, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Chronic rhinosinusitis without nasal polyps (CRSsNP) or Chronic rhinosinusitis with nasal polyps (CRSwNP).

Exclusion Criteria:

* Patients with significant nasal polyps (as determined by a clinician) were excluded upfront due to the unlikeness of irrigation penetration regardless of the head position. Patients with significant atopy, cystic fibrosis, granulomatosis with polyangiitis or other connective tissue disorder, and current pregnancy were also excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2027-06-26 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Nasal Obstruction Symptom Evaluation (NOSE) score | completed at baseline and after 8 weeks of treatment.
  patient-reported outcome measure
22-item Sino-Nasal Outcome Test (SNOT-22) score | completed at baseline and after 8 weeks of treatment.
  patient-reported outcome measure
Visual Analogue Scale (VAS) of nasal congestion score | completed at baseline and after 8 weeks of treatment.
  patient-reported outcome measure
Lund-Mackay (LM) score of sinus inflammation. | assessed from CT scans taken at baseline and after 8 weeks of treatment.
  Objective rating of sinus inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Eye and Ear Institue, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Albu S. Chronic Rhinosinusitis-An Update on Epidemiology, Pathogenesis and Management. J Clin Med. 2020 Jul 18;9(7):2285. doi: 10.3390/jcm9072285. PMID 32708447
- [Background] Wormald PJ, Cain T, Oates L, Hawke L, Wong I. A comparative study of three methods of nasal irrigation. Laryngoscope. 2004 Dec;114(12):2224-7. doi: 10.1097/01.mlg.0000149463.95950.c5. PMID 15564850
- [Background] Piromchai P, Puvatanond C, Kirtsreesakul V, Chaiyasate S, Suwanwech T. A multicenter survey on the effectiveness of nasal irrigation devices in rhinosinusitis patients. Laryngoscope Investig Otolaryngol. 2020 Nov 16;5(6):1003-1010. doi: 10.1002/lio2.497. eCollection 2020 Dec. PMID 33364388
- [Background] Lepley TJ, Kim K, Ardizzone M, Kelly KM, Otto BA, Zhao K. 3D Printing as a Planning Tool to Optimize Sinonasal Irrigation. Ann Otol Rhinol Laryngol. 2023 Nov;132(11):1306-1313. doi: 10.1177/00034894221149242. Epub 2023 Jan 26. PMID 36704822
- [Background] Zhao K, Kim K, Craig JR, Palmer JN. Using 3D printed sinonasal models to visualize and optimize personalized sinonasal sinus irrigation strategies. Rhinology. 2020 Jun 1;58(3):266-272. doi: 10.4193/Rhin19.314. PMID 32441708
- [Derived] Root ZT, Lepley TJ, Kim K, Schneller AR, Zhao S, Wen R, Formanek VL, Sussman SM, Lee JS, Odeh A, Wei L, Kelly KM, Otto BA, Zhao K. Optimizing Corticosteroid Sinonasal Irrigation Outcomes Through 3D Printing: A Randomized Pilot Clinical Trial. OTO Open. 2024 Oct 16;8(4):e70036. doi: 10.1002/oto2.70036. eCollection 2024 Oct-Dec. PMID 39417152